CLINICAL TRIAL: NCT01281631
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of NP001 in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study of NP001 in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuraltus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP001-10-002
Record Dates: First submitted 2011-01-17; First posted 2011-01-24 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose NP001 (Experimental): Low drug dose
  Interventions: Drug: NP001
- High dose NP001 (Experimental): High drug dose
  Interventions: Drug: NP001
- Placebo (Placebo Comparator): normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NP001 — Low dose of NP001
  Arms: Low dose NP001
Drug: NP001 — High dose of NP001
  Arms: High dose NP001
Drug: Placebo — normal saline
  Arms: Placebo

SUMMARY:
This is a Phase 2 randomized, double-blind, placebo-controlled, multicenter study of NP001 in subjects with ALS.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study of NP001 in subjects with ALS conducted in multiple centers. Drug or placebo will be given intravenously. Approximately 105 subjects will be enrolled. Subjects will be allocated (1:1:1) to placebo and 2 dose levels of NP001.

ELIGIBILITY:
Subjects with sporadic or familial ALS classified as definite, probable, or laboratory-supported probable ALS according to the revised El Escorial criteria. A list of key criteria is listed below:

Inclusion Criteria:

* Onset of symptoms less than 3 years prior to study entry.
* Forced Vital Capacity (FVC) at least 70% of that predicted for age and height.
* Stable dose of riluzole if undergoing treatment with this agent.
* For females: Not be of childbearing potential or agree to use adequate birth control during the study.

Exclusion Criteria:

* Unstable medical condition(s) other than ALS.
* Life expectancy of less than 6 months.
* Require life-sustaining interventions for the 6 months following randomization.
* Have a tracheotomy or be using ventilatory assistance [including Bi-level Positive Airway Pressure (BiPAP) or Continuous Positive Airway Pressure (CPAP)].
* Active pulmonary disease.
* Immune modulator therapy within 12 weeks of study entry or participation in studies of other agents within the last 4 weeks prior to the randomization.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of NP001 on measures of clinical function | over 9 months

SECONDARY OUTCOMES:
Safety and tolerability in ALS | duration of study
Pulmonary function and biomarkers | over 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert G. Miller, MD, Principal Investigator — Forbes Norris ALS Treatment and Research, California Pacific Medical Center
Locations (17):
- United States (17):
  - Mayo Clinic, Scottsdale, Scottsdale, Arizona
  - UC, Irvine, Irvine, California
  - UCLA, Los Angeles, California
  - California Pacific Med Center Forbes Norris MDA/ALS Research and Treatment Center, San Francisco, California
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - The Emory Clinic, Atlanta, Georgia
  - University of Kansas Medical Center, Landon Center on Aging, Kansas City, Kansas
  - University of Kentucky, Department of Neurology, Lexington, Kentucky
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Columbia University, New York, New York
  - SUNY Upstate Medical University, Syracuse, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Dept of Neurology, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Providence ALS Center, Portland, Oregon
  - Methodist Hospital Research Institute, Methodist Neurologic Institute, Houston, Texas
  - Providence Saint Peter Hospital, Centralia, Washington

REFERENCES:
- [Derived] Forrest BD, Goyal NA, Fleming TR, Bracci PM, Brett NR, Khan Z, Robinson M, Azhir A, McGrath M. The Effectiveness of NP001 on the Long-Term Survival of Patients with Amyotrophic Lateral Sclerosis. Biomedicines. 2024 Oct 16;12(10):2367. doi: 10.3390/biomedicines12102367. PMID 39457678